CLINICAL TRIAL: NCT06600334
Title: Prevalence of Osteoporosis Among Inflammatory Bowel Disease Patients in Assiut University Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Dina Fathy (Other)
Responsible Party: Sponsor-Investigator, Dina Fathy, Dina Fathy, Assiut University
Organization: Assiut University (Other)
Other Study IDs: osteoporosis and IBD patients
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Osteoporosis
Keywords: Prevalence of osteoporosis among inflammatory bowel disease patients in Assiut university hospitals.
MeSH Terms: conditions — Osteoporosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: dexa scan — Bone density scans

SUMMARY:
the prevalence of osteoporosis in patients with inflammatory bowel disease in Assiut University Hospitals.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) includes ulcerative colitis (UC) and Crohn's disease (CD) (1) .There has been a global rise in the incidence of IBD over the last few decades. (2) In the course of this disease, apart from the involvement of the gastrointestinal tract, up to 50% of patients may also have extraintestinal manifestations (EIMs) .One of them may be osteoporosis (OST), which is present in over half of IBD patients; this constitutes a significant problem due to the increased risk of fractures, especially non-traumatic fractures.(3) Known risk factors for OST in IBD include the persistence of chronic inflammation, treatment with glucocorticosteroids, extensive range of the disease, previous resection of the small intestine, arthralgia, and current nutritional deficiencies. Some risk factors are similar to those found in the general population, such as age, smoking, or low physical activity.(3) The pathogenesis of osteoporosis is multifactorial and comprises such elements as steroid therapy, low body mass index (BMI), malnutrition, genetic predispositions, and vitamin D deficiency (4) Given that the gastroenterologist is often regarded as the main provider for IBD patients, gastroenterologists and primary care physicians are equally responsible to recommend preventive measures and screening for osteoporosis, in addition to other healthcare maintenance issues.(5) Dual energy X-ray absorptiometry (DEXA) scans are globally recognised as the screening tool for low BMD (6) The Z and T scores are used to establish the diagnosis of osteoporosis, osteopenia or low BMD according to the 2019 International Society of Clinical Densitometry official position for adults.(7)

ELIGIBILITY:
Inclusion Criteria:

* The study will include Patients aged 18-65 years, diagnosed with either Crohn's disease or ulcerative colitis, The diagnosis of UC and CD based on the clinical, endoscopic, laboratory and histological criteria according to ECCO Guidelines. The activity of IBD will be determined with the use of the Crohn's Disease Activity Index (CDAI) for CD, and the Mayo score for UC, data collection will obtained over one year duration

Exclusion Criteria:

1. Patients Known to have osteoporosis and on treatment
2. Female patients on COCs
3. Patients with malignancy
4. Patients with CKD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cases of IBD in Internal medicine department, Assiut University Hospitals.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
1- To detect the prevalence of osteoporosis in patients with inflammatory bowel disease in Assiut University Hospitals. | 1 year

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lewandowski K, Kaniewska M, Wiecek M, Szwarc P, Panufnik P, Tulewicz-Marti E, Walicka M, Franek E, Rydzewska G. Risk Factors for Osteoporosis among Patients with Inflammatory Bowel Disease-Do We Already Know Everything? Nutrients. 2023 Feb 24;15(5):1151. doi: 10.3390/nu15051151. PMID 36904150
- [Result] Frisoli A Jr, Paes AT, Kimura AD, Azevedo E, Ambrosio V. Measuring forearm bone density instead of lumbar spine bone density improves the sensitivity of diagnosing osteoporosis in older adults with cardiovascular diseases: Data from SARCOS study. Bone Rep. 2021 Oct 4;15:101134. doi: 10.1016/j.bonr.2021.101134. eCollection 2021 Dec. PMID 34660851